CLINICAL TRIAL: NCT00466752
Title: A Phase II Study of Sorafenib (Nexavar®) Prior to Radical Prostatectomy in Patients With High-Risk Localized Prostate Cancer
Brief Title: Sorafenib Tosylate and Gene Expression Analysis in Patients Undergoing Surgery For High-Risk Localized Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Evan Y. Yu, MD, Principal Investigator, University of Washington
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 6307; NCI-2010-00604 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2007-04-25; First posted 2007-04-27 (Estimated); Results first posted 2017-11-22 (Actual); Last update posted 2017-11-22 (Actual); Status verified 2017-11

CONDITIONS: Adenocarcinoma of the Prostate; Stage II Prostate Cancer; Stage III Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Sorafenib; Microarray Analysis; Gene Expression Profiling; Immunohistochemistry; Biopsy, Needle; Blotting, Western

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment (enzyme inhibitor) 48hr stop (Experimental): Patients receive sorafenib tosylate PO BID on days 1-14. Treatment repeats every 2 weeks for 3 courses in the absence of disease progression or unacceptable toxicity. Beginning 2 days after completion of sorafenib tosylate, patients undergo radical prostatectomy on approximately day 43.
  Interventions: Drug: sorafenib tosylate; Genetic: microarray analysis; Other: immunohistochemistry staining method; Genetic: gene expression analysis; Procedure: needle biopsy; Procedure: therapeutic conventional surgery; Other: laboratory biomarker analysis; Genetic: western blotting; Genetic: RNA analysis
- Treatment (enzyme inhibitor) 24hr stop (Experimental): tients receive sorafenib tosylate PO BID on days 1-14. Treatment repeats every 2 weeks for 3 courses in the absence of disease progression or unacceptable toxicity. Beginning 1 day after completion of sorafenib tosylate, patients undergo radical prostatectomy on approximately day 43.
  Interventions: Drug: sorafenib tosylate; Genetic: microarray analysis; Other: immunohistochemistry staining method; Genetic: gene expression analysis; Procedure: needle biopsy; Procedure: therapeutic conventional surgery; Other: laboratory biomarker analysis; Genetic: western blotting; Genetic: RNA analysis

INTERVENTIONS:
Drug: sorafenib tosylate — Given PO
  Other Names: BAY 43-9006; BAY 43-9006 Tosylate Salt; BAY 54-9085; Nexavar; SFN
Genetic: microarray analysis — Correlative studies
  Other Names: gene expression profiling
Other: immunohistochemistry staining method — Correlative studies
  Other Names: immunohistochemistry
Genetic: gene expression analysis — Correlative studies
Procedure: needle biopsy — Correlative studies
  Other Names: aspiration biopsy; puncture biopsy
Procedure: therapeutic conventional surgery — Undergo prostatectomy
Other: laboratory biomarker analysis — Correlative studies
Genetic: western blotting — Correlative studies
  Other Names: Blotting, Western; Western Blot
Genetic: RNA analysis — Correlative studies

SUMMARY:
This phase II trial is studying sorafenib tosylate and gene expression in patients undergoing surgery for high-risk localized prostate cancer. Sorafenib tosylate may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor. Studying samples of blood and tumor tissues in the laboratory from patients with prostate cancer may help doctors learn more about changes that occur in DNA after treatment with sorafenib tosylate

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To compare the gene expression changes (transcript profiles) between pre- and post-treatment tumor specimens in order to determine the molecular impact of multi-kinase inhibition on prostate cancer. While this analysis will initially be targeted to tumor cells, gene expression changes in the surrounding stromal tissue may also be analyzed.

SECONDARY OBJECTIVES:

I. To determine if specific downstream protein effectors (i.e. ERK, AKT, and S6- kinase) of Sorafenib kinase targets are affected by changes in protein phosphorylation by immunohistochemistry.

II. To provide evidence that Sorafenib has significant anti-tumor effect by comparison of pre- and post-treatment immunohistochemical markers of apoptosis (caspase-3), cell proliferation (Ki-67), and angiogenesis (microvessel density).

III. To determine the pathologic complete response rate, defined as absence of cancer in the prostatectomy specimen.

IV. To determine rates of positive surgical margins, extracapsular extension, seminal vesicle and lymph node involvement with tumor in comparison with Memorial Sloan Kettering pre-operative nomogram predictions.

V. To determine the percentage of patients with a >= 25% and >= 50% decline in PSA while receiving Sorafenib.

VI. To determine tissue Sorafenib levels in prostate tumors after treatment and correlate with molecular, clinical, and/or pathologic outcomes.

VII. To describe changes in overall histology after treatment with Sorafenib and correlate with molecular and clinical outcomes.

VIII. To determine if patients with baseline alterations in phospho-ERK, phospho-AKT, and phospho-S6-kinase expression correlate with treatment related molecular, clinical, and/or pathologic outcomes.

IX. To collect tissue samples for future analysis of correlative biomarkers of prognosis or treatment response.

X. To collect frozen plasma for future analysis of correlative biomarkers of treatment response (no genetic analysis will be performed on these specimens).

OUTLINE:

Patients receive sorafenib tosylate orally (PO) twice daily (BID) on days 1-14. Treatment repeats every 2 weeks for 3 courses in the absence of disease progression or unacceptable toxicity. Beginning 1 or 2 days after completion of sorafenib tosylate, patients undergo radical prostatectomy on approximately day 43.

After completion of study treatment, patients are followed up for 6-10 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of the prostate
* Radical prostatectomy and lymph node dissection planned as primary therapy in a patient with acceptable surgical risk (e.g., cardiovascular, pulmonary, and functional status)
* 10 year or longer life expectancy
* Any of the following high-risk features: Clinical stage T2b (palpable bilateral involvement) OR surgically resectable T3 OR PSA >= 20 ng/ml OR overall Gleason grade >= 8
* No evidence of bone metastases on bone scan
* No evidence of lymph nodes >= 2 cm in diameter on pelvic CT scan
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2
* Hemoglobin >= 9.0 g/dl
* Absolute neutrophil count (ANC) >= 1,500/mm^3
* Platelet count >= 100,000/mm^3
* Total bilirubin =< 1.5 x ULN
* ALT =< 2.5 x the ULN
* AST =< 2.5 x the ULN
* INR =< 1.5 and aPTT within normal limits
* Creatinine =< 1.5 x ULN or creatinine clearance > 60mL/min/1.73 m^2
* Men must agree to use adequate contraception (abstinence, hormonal in female partner, or barrier method of birth control) prior to study entry, for the duration of study participation, and for at least two weeks after stopping treatment
* Signed informed patient consent

Exclusion Criteria:

* Prior therapy for prostate cancer including conventional androgen deprivation therapy, radiotherapy (external beam or brachytherapy), cryotherapy, and/or cytotoxic chemotherapy
* Any known metastasis; patients with neurological symptoms must undergo a CT scan/MRI of the brain to exclude brain metastasis
* Significant active medical illness which in the opinion of the investigator would preclude protocol treatment
* Another malignancy, other than non-melanoma skin cancer, during the past 5 years
* History of bleeding diathesis or unexpected surgical bleeding
* Patients with active coagulopathy
* Cardiac disease: Congestive heart failure > class II NYHA; patients must not have unstable angina (anginal symptoms at rest) or new onset angina (began within the last 3 months) or myocardial infarction within the past 6 months
* Cardiac ventricular arrhythmias requiring anti-arrhythmic therapy
* Uncontrolled hypertension, as defined by systolic blood pressure consistently in excess of 150 mmHg, or diastolic pressure consistently in excess of 90 mmHg
* Thrombolic or embolic events such as a cerebrovascular accident including transient ischemic attacks within the past 6 months
* Pulmonary hemorrhage/bleeding event >= CTCAE Grade 2 within 4 weeks of first dose of study drug
* Any other hemorrhage/bleeding event >= CTCAE Grade 3 within 4 weeks of first dose of study drug
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to sorafenib
* Patients may not be concurrently receiving any chemotherapy, immunotherapy, hormonal therapy, or molecular targeted agents to treat their prostate cancer
* Patients may not be receiving any other investigational agents
* Therapeutic anticoagulation with heparin, low-molecular weight heparin, or warfarin within the last 4 weeks
* Patients may not be using rifampin, digoxin, quinidine, ketoconazole, itraconazole, cyclosporine, carbamazepine, phenytoin, phenobarbital, St. John's Wart, or products containing grapefruit juice
* Patients may not be using bevacizumab or any other drugs that target VEGF or VEGF receptors
* Active clinically significant infections (>= grade 2 NCI-CTCAE version 3.0); patients may enroll after infection resolves
* HIV-positive patients receiving combination anti-retroviral therapy because of possible pharmacokinetic interactions with Sorafenib
* Any condition that impairs patient's ability to swallow whole pills
* Any malabsorption problem

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2006-12; Primary Completion 2010-04 (Actual); Study Completion 2011-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Evan Yu, Principal Investigator — Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Locations (1):
- Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were screened and enrolled at a single site in Seattle, Washington, United States.
Pre-assignment Details: Five subjects were screened for this study, deemed eligible and enrolled.
Groups:
- 48 Hour Drug Stop Point: Sorafenib 400mg taken orally twice per day for 41 days prior to radical prostatectomy. Last dose of study drug is the morning dose 2 days prior to surgery.
- 24 Hour Drug Stop Point: Sorafenib 400mg taken orally twice per day for 42 days prior to radical prostatectomy. Last dose of study drug is the morning dose the day prior to surgery.
Period: Overall Study
Arm/Group | 48 Hour Drug Stop Point | 24 Hour Drug Stop Point
Started | 5 | 0
Completed | 5 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 48 Hour Drug Stop Point | 24 Hour Drug Stop Point | Total
Number analyzed (Participants) | 5 | 0 | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 0 | 4
  >=65 years | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 5 | 0 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 4 | 0 | 4
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 5 | 0 | 5
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 5 |  | 5
Baseline PSA [Median (Full Range); unit: ng/mL] | 14.76 [6.14 to 120.76] |  | 14.76 [6.14 to 120.76]
Gleason Score at Diagnosis [Median (Full Range); unit: units on a scale] — Gleason score is the sum of 2 numbers,each between 1-5, representing the pattern of tumor cells seen by a pathologist reviewing a prostate biopsy. 1 is given to cells that resemble normal cells. 5 is given to cells that least resemble normal cells. 1st number represents the most predominant cell pattern in a prostate biopsy, 2nd number represents the 2nd most predominant cell pattern in the same biopsy. Gleason score is the sum of these numbers. Lower Gleason scores (2-4) have been associated with less aggressive cancers, higher Gleason scores have been associated with more aggressive cancers.
  units on a scale | 7 [7 to 9] |  | 7 [7 to 9]

OUTCOME MEASURES:

1. Primary Outcome: Efficacy as Assessed by Number of Patients With Changes Across Transcript Profiles by Microarray Analysis in Prostate Cancer Specimens, Specifically Those With Complete Pathologic Response.
Description: Determined by changes across transcript profiles, by microarray analysis, in pre- versus post-treatment prostate cancer specimens (minimum 50 day time frame between these). Proportion of patients with complete pathologic response.
Time Frame: Pre- versus post-treatment
Population: Data not collected
Arm/Group | 48 Hour Drug Stop Point | 24 Hour Drug Stop Point
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Number of Participants With Complete Pathologic Response
Description: Proportion of Patients with at least 50% decline in PSA on Day 1 of Cycle 2, Day 1 of Cycle 3, and on day of radical prostatectomy.
Time Frame: Day 1 of cycles 2 and 3, and day of radical prostatectomy. Each cycle is 2 weeks.
Population: One patient did not have lab samples collected on day of radical prostatectomy.
Measure: Count of Participants; unit: Participants
Arm/Group | 48 Hour Drug Stop Point | 24 Hour Drug Stop Point
Number analyzed (Participants) | 5 | 0
Participants
  Day 1 of Cycle 2 | 0 |
  Day 1 of Cycle 3 | 0 |
  Day of Radical Prostatectomy: number analyzed (Participants) | 4 | 0
  Day of Radical Prostatectomy | 0 |

3. Secondary Outcome: Number of Participants With at Least 25% Reduction in PSA
Description: Proportion of Patients with at least 25% decline in PSA on Day 1 of Cycle 2, Day 1 of Cycle 3, and on day of radical prostatectomy.
Time Frame: Day 1 of cycles 2 and 3 and on the day of radical prostatectomy. Each cycle is 2 weeks.
Population: One patient did not have lab samples collected on day of radical prostatectomy.
Measure: Count of Participants; unit: Participants
Arm/Group | 48 Hour Drug Stop Point | 24 Hour Drug Stop Point
Number analyzed (Participants) | 5 | 0
Participants
  Day 1 of Cycle 2 | 0 |
  Day 1 of Cycle 3 | 0 |
  Day of Radical Prostatectomy: number analyzed (Participants) | 4 | 0
  Day of Radical Prostatectomy | 1 |

ADVERSE EVENTS:
Time Frame: Reported Adverse Events (AEs) include events starting on or after Day 0 and on or before Day 113
Description: If a subject experienced more than 1 of a given AE, the subject is counted only once for that AE.
Arm/Group | 48 Hour Drug Stop Point | 24 Hour Drug Stop Point
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/0
Other Adverse Events (participants affected / at risk) | 5/5 | 0/0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 48 Hour Drug Stop Point (N=5) | 24 Hour Drug Stop Point (N=0)
Tinnitus (Ear and labyrinth disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 2 | 0
pain, gastrointestinal, oral cavity, esophagus (General disorders) | 1 | 0
pain, renal/genitourinary (General disorders) | 1 | 0
Fatigue (General disorders) | 3 | 0
Weight loss (General disorders) | 1 | 0
Pancreatitis (Hepatobiliary disorders) | 1 | 0
Transaminitis (Metabolism and nutrition disorders) | 1 | 0
pain, musculoskeletal, extremity-limb (Musculoskeletal and connective tissue disorders) | 1 | 0
Tingling feet and scalp (Nervous system disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0
urination frequency and urgency (Renal and urinary disorders) | 1 | 0
Gynecomastia (Reproductive system and breast disorders) | 1 | 0
voice changes/dysarthria (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0
Hand-foot syndrome (Skin and subcutaneous tissue disorders) | 2 | 0
Pruritis (Skin and subcutaneous tissue disorders) | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 0
Hypertension (Vascular disorders) | 4 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes